CLINICAL TRIAL: NCT04758767
Title: A Phase 1 Dose Escalation and Expansion Study of CID-103, an Anti-CD38 Antibody, in Patients With Previously Treated Relapsed or Refractory Multiple Myeloma
Brief Title: CID-103 (Anti-CD38 Antibody) in Previously Treated Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CASI-CID-103-101; 2019-004006-10 (EudraCT Number)
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; CID-103; anti-CD38 antibody
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Single arm dose escalation, followed by dose expansion arm (2 cohorts)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation cohort (Experimental): Monotherapy CID-103. Priming dose will be given for first dose. Dose and duration of infusion dependent on dose cohort and tolerability.
  Interventions: Drug: CID-103
- Dose expansion cohort - pretreated (Experimental): CID-103 monotherapy at the recommended phase 2 dose
  Interventions: Drug: CID-103
- Dose expansion cohort - Naïve (Experimental): CID-103 monotherapy at the recommended phase 2 dose
  Interventions: Drug: CID-103

INTERVENTIONS:
Drug: CID-103 — anti-CD38 antibody

SUMMARY:
Patients with relapsed/refractory multiple myeloma will be enrolled in a dose-escalation phase receiving monotherapy CID-103. Once the recommended CID-103 dose and infusion duration is known, additional patients will be enrolled in an expansion phase consisting of two cohorts (anti-CD38 pretreated, and anti-CD38 treatment naïve). Patients will be treated until disease progression or unacceptable toxicities.

DETAILED DESCRIPTION:
Dose escalation/infusion duration phase:

During the CID-103 dose escalation/infusion duration phase, only patients diagnosed with multiple myeloma who have relapsed or are refractory to at least two prior lines of therapy including a proteasome inhibitor, an immunomodulatory agent and an anti-CD38 antibody will be enrolled. Patients will receive monotherapy CID-103. Dose escalation decisions will be based on dose-limiting toxicities; infusion duration decisions will be based on infusion-related reactions. The dose taken forward into the expansion phase will be the RP2D determined in the dose escalation phase.

Expansion phase:

The expansion phase consists of two specific cohorts of patients with relapsed/refractory multiple myeloma: 1) Pretreated cohort having received previous treatment with an anti-CD38 antibody and 2) Naïve cohort in patients for whom an anti-CD38 antibody is unavailable. Eight patients will be enrolled into each cohort, and if one or more responses is observed, that cohort will be expanded to a total of 14 patients to further assess efficacy. Patients must have had at least two prior systemic therapies (mono or combo), including a proteasome inhibitor and an immunomodulatory agent. Patients will be treated until disease progression or unacceptable toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to sign the ICF and comply with the protocol
2. Male or female ≥ 18 years of age
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
4. Agrees to bone marrow aspirates
5. Must have pathologically confirmed multiple myeloma
6. Has relapsed or refractory myeloma
7. At least 2 prior systemic anti-cancer therapies for relapsed or refractory multiple myeloma, including an immunomodulatory agent and a proteasome inhibitor
8. Meets all IMWG 2014 criteria at diagnosis or at time of current relapse
9. Measurable disease
10. If female, must be of non-childbearing potential, or have a negative pregnancy test at screening and use highly adequate contraception throughout study until 90 days after last dose
11. If male with partner of childbearing potential, be vasectomized or female partner must use highly adequate contraception throughout study until 180 days after last dose
12. All previous therapy-related adverse events should have resolved, prior to Day 1, to Grade 1 or baseline value with the exception of alopecia (includes effects of radiotherapy)
13. Adequate organ function as indicated by neutrophils, platelets, hemoglobin, eGFR, serum total and direct bilirubin, AST, ALT, INR, aPTT

Exclusion Criteria:

1. Received small molecule or tyrosine kinase inhibitor within two weeks or five half-lives (whichever is longer) prior to the first dose of study drug; chemotherapy or biological cell-based cancer therapy within four weeks prior to the first dose of study drug; nitrosourea or radioisotope within six weeks prior to first dose of study drug, non-recovery to the CTCAE v5 Grade 1 or better from the adverse events due to cancer therapeutics administered more than four weeks earlier.
2. Received an anti-CD38 therapy within four months from first dose of study drug
3. Inability to perform study baseline RBC type and cross-match, phenotype, genotype (if applicable) or lack of available baseline data on RBC phenotype or genotype (if applicable)
4. Receiving other concurrent investigational therapies or have received investigational therapies within four weeks of the first dose of study drug or five half-lives, if known, whichever is shorter
5. Currently receiving systemic steroids unless equivalent to 10 mg/day of prednisone or less for adrenal replacement only. At least two weeks since last dose of steroid therapy intended for the treatment of myeloma and the first dose of study drug.
6. Non-secretory myeloma unless measurable plasmacytoma
7. Known hypersensitivity to CID-103 excipients or prior severe hypersensitivity to a monoclonal antibody
8. Baseline interval between Q and T wave on electrocardiogram > 480 msec using Fridericia's formula (QTcF)
9. Requires renal dialysis
10. Sensory or motor neuropathy ≥ Grade 3
11. Known/clinically significant amyloidosis
12. Known active central nervous system disease or leptomeningeal plasmacytoma.
13. Presence of any other active malignancy requiring systemic therapy other than the disease under study
14. Active infection requiring systemic therapy
15. Active infection with human immunodeficiency virus and CD4+ T-cell count < 350/μL
16. Active infection with hepatitis B (surface antigen); or infection with hepatitis C in absence of sustained virologic response
17. Therapeutic anticoagulation, meaning any thromboembolic event within the last six months prior to first dose of study drug or anticoagulation with therapeutic (non-prophylactic) intent
18. A history or evidence of cardiovascular risk
19. History or clinical evidence of any surgical or medical condition which the investigator judges as likely to interfere with the results of the study or pose an additional risk in participating, particularly any pre-existing condition that would put the patient at additional risk should they experience an infusion-related reaction
20. At the time of signing informed consent is a regular user (including "recreational/medical use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Adverse events | approximately 18 months after study start
  CTCAE v5 coded using the current Medical Dictionary for Regulatory Activities (MedDRA) version

SECONDARY OUTCOMES:
Recommended Phase 2 dose | approximately 18 months after study start
  Based primarily on dose-limiting toxicities
Optimal pre- and post-medication regimens | approximately 18 months after study start
  Type, incidence, severity, timing, seriousness, and relatedness of AEs and laboratory abnormalities will be compared before and after the changes in pre/post medications are made, with specific focus on IRRs and their symptoms
Target engagement assays and ex vivo testing | approximately 18 months after study start
  Extent of RBC binding and cross-match confounding
PK - AUC of CID-103 | approximately 18 months and 3 years after study start
  AUC of CID-103 in serum
PK - Cmax of CID-103 | approximately 18 months and 3 years after study start
  Cmax of CID-103 in serum
PK - t1/2 of CID-103 | approximately 18 months and 3 years after study start
  half-life of CID-103 in serum
PK - Vd of CID-103 | approximately 18 months and 3 years after study start
  volume of distribution of CID-103 in serum
PK - accumulation of CID-103 | approximately 18 months and 3 years after study start
  accumulation of CID-103 in serum
Objective response rate | approximately 3 years after study start
  Based on IMWG
Duration of response | approximately 3 years after study start
  Calculated using a Kaplan-Meier method overall and for appropriate subgroups and cohorts, based on IMWG
Progression-free survival | approximately 3 years after study start
  Calculated using a Kaplan-Meier method overall and for appropriate subgroups and cohorts, based on IMWG
Overall survival | approximately 3 years after study start
  Calculated using a Kaplan-Meier method overall and for appropriate subgroups and cohorts, based on IMWG

OTHER OUTCOMES:
Target binding of CID-103 | approximately 3 years after study start
  Target binding on different circulating blood cell populations and the potential PD markers

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zukiwski, MD, Study Director — CASI Pharmaceuticals, Inc.
Locations (4):
- France (3):
  - CHU de Nantes - Hôpital Hôtel-Dieu, Nantes
  - CHU Rennes - Pontchaillou, Rennes
  - Gustave Roussy Cancer Center, Villejuif
- Sarah Cannon, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No